CLINICAL TRIAL: NCT02054988
Title: "Potential Effect of Acute and Chronic Caffeine Administration on Platelet Reactivity in Patient With Coronary Artery Disease on Dual Antiplatelet Therapy"
Acronym: CyCLOPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Polacco Marina, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: PM3110
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: CORONARY ARTERY DISEASE
MeSH Terms: conditions — Coronary Artery Disease | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- caffeine (Experimental): three cups of coffee will be administered for 10 days (on chronic phase) and two cups of coffee will be consecutively administered for "acute" evaluation.
  Interventions: Other: caffeine
- not caffeine (Active Comparator): not caffeine will be administered for the duration of the study
  Interventions: Other: not caffeine

INTERVENTIONS:
Other: caffeine — After 5 day coffee wash-out period, patients were randomly assigned to caffeine for 10 days. At baseline: 2 cups of coffee consecutively after 5 hour by clopidogrel or prasugrel intake. Afterwards, 3 cups of coffee daily for 10 days.
  Platelet reactivity (expressed as P2Y(12) reaction units (PRU) by the point-of-care VerifyNow assay [Accumetrics, San Diego, California]) was measured at baseline and after 10-days of coffee intake.
  Arms: caffeine
Other: not caffeine — evaluate the platelet reactivity after 10 days of no caffeine intake
  Arms: not caffeine

SUMMARY:
Prasugrel is a potent thienopyridine antiplatelet agent that selectively and irreversibly inhibits ADP-induced platelet aggregation mediated by the P2Y12 receptor. Prasugrel is a prodrug that must first undergo biotransformation to its active metabolite via cytochrome P450-mediated hepatic metabolism (CYP1A2). Clopidogrel is currently administered to several million patients especially after coronary stenting. Clopidogrel has been shown to reduce cardiovascular complications in patients with acute coronary syndromes and patients who have undergone coronary stenting. The mechanism of action of clopidogrel's active metabolite involves inhibition of the purinergic adenosine diphosphate (ADP) receptor P2Y12 on the platelet membrane. Blockade of this receptor prevents uncoupling of the associated Gi2 protein which ultimately leads to increased platelet cyclic AMP (cAMP) formation.3 Cyclic AMP is a key signaling molecule in inhibiting platelet aggregation, but its intracellular levels are affected by several other commonly used compounds. For instance, methylxanthines, such as caffeine, theophylline, and theobromine (an ingredient of chocolate), all cause elevation of intracellular cAMP levels by inhibiting adenosine receptors (types A1 and A2) on the platelet membrane. The effect of caffeine consumption on platelet reactivity depends on the caffeine dose and duration of administration. Chronic caffeine consumption (≥7 days) appears to be associated with inhibition of platelet aggregation, probably through upregulation of adenosine receptors.The aim of this study was to examine the effect of acute caffeine consumption, at a dose equivalent to commercial coffee drinks, on the antiplatelet effect of clopidogrel and prasugrel, in patients with coronary artery disease (CAD).

Platelet function will be evaluated using a validated method: the VerifyNow System (Accumetrics Inc., San Diego, CA), which is a point-of-care turbidimetry-based optical detection system that measures platelet-induced aggregation.

DETAILED DESCRIPTION:
Prasugrel is a potent thienopyridine antiplatelet agent that selectively and irreversibly inhibits ADP-induced platelet aggregation mediated by the P2Y12 receptor. Prasugrel is a prodrug that must first undergo biotransformation to its active metabolite via cytochrome P450-mediated hepatic metabolism (CYP1A2). Clopidogrel is currently administered to several million patients especially after coronary stenting. Clopidogrel has been shown to reduce cardiovascular complications in patients with acute coronary syndromes and patients who have undergone coronary stenting. The mechanism of action of clopidogrel's active metabolite involves inhibition of the purinergic adenosine diphosphate (ADP) receptor P2Y12 on the platelet membrane. Blockade of this receptor prevents uncoupling of the associated Gi2 protein which ultimately leads to increased platelet cyclic AMP (cAMP) formation.3 Cyclic AMP is a key signaling molecule in inhibiting platelet aggregation, but its intracellular levels are affected by several other commonly used compounds. For instance, methylxanthines, such as caffeine, theophylline, and theobromine (an ingredient of chocolate), all cause elevation of intracellular cAMP levels by inhibiting adenosine receptors (types A1 and A2) on the platelet membrane. The effect of caffeine consumption on platelet reactivity depends on the caffeine dose and duration of administration. Chronic caffeine consumption (≥7 days) appears to be associated with inhibition of platelet aggregation, probably through upregulation of adenosine receptors. The effect of acute caffeine administration on platelet function is less clear. Different studies have shown either an increase, decrease, or no change in platelet reactivity after acute caffeine administration. The aim of this study was to examine the effect of acute caffeine consumption, at a dose equivalent to commercial coffee drinks, on the antiplatelet effect of clopidogrel and prasugrel, in patients with coronary artery disease (CAD).

Platelet function will be evaluated using a validated method: the VerifyNow System (Accumetrics Inc., San Diego, CA), which is a point-of-care turbidimetry-based optical detection system that measures platelet-induced aggregation. Platelet function will be measured with the VerifyNow P2Y12 test at baseline, (after 5 day wash-out period to avoid any carryover effect ) and after 10 days of taking caffeine.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients undergone PTCA
2. Patients on dual antiplatelet therapy with ASA and clopidogrel or prasugrel or ticagrelor.

Exclusion Criteria:

1. People unable to understand and willing to sign the informed consent form;
2. Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units | After 10 days of caffeine intake
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California]

CONTACTS AND LOCATIONS:
Overall Officials: Marina MD Polacco, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Rome, Lazio, Italy